CLINICAL TRIAL: NCT01566682
Title: A Multi-Center Trial of the ProLung Test™ (Transthoracic Bioconductance Measurement) as an Adjunct to CT Chest Scans for the Risk Stratification of Patients With Pulmonary Lesions Suspicious for Lung Cancer
Brief Title: A Multi-Center Trial of the ProLung Test™
Status: Completed | Type: Observational
Sponsor: Fresh Medical Laboratories (Industry)
Collaborators: Huntsman Cancer Institute (Other); University of California, Los Angeles (Other); Henry Ford Health System (Other); University of California, San Diego (Other); Intermountain Health Care, Inc. (Other); M.D. Anderson Cancer Center (Other); Greater Baltimore Medical Center (Other); Stanford University (Other); Loyola University (Other); Providence Health Center (Unknown); Wake Forest (Unknown); University of Minnesota Masonic Cancer Center (Unknown); Beth Israel Deaconess Medical Center (Other); Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: PL-208
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Solitary Pulmonary Nodule; Multiple Pulmonary Nodules
Keywords: Lung Lesion; Lung Mass; Lung Nodule; Lung Cancer; Low-Dose CT; CT; Diagnostic; Evaluation; Bioconductance; ProLung
MeSH Terms: conditions — Solitary Pulmonary Nodule; Multiple Pulmonary Nodules; Lung Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Indeterminate Pulmonary Lesions: Patients with Pulmonary Lesions as seen by CT

SUMMARY:
The primary Study hypothesis is that the ProLung Test will demonstrate safety and efficacy in the risk stratification of patients with pulmonary lesions identified by CT that are suspicious for lung cancer. A statistically significant result will indicate that patients with a high ProLung Test result have a greater risk of developing lung cancer than patients with a low test result.

There are three Specific Aims of this study:

1. Optimize and confirm the stability of the ProLung Test risk-stratification algorithm in patients with a diagnosis.
2. Externally validate the efficacy of the ProLung Test risk-stratification algorithm by comparing the test result to the conclusive patient diagnosis.
3. Assess the safety and tolerability of the ProLung Test procedures.

Study Design This Study consists of two distinct phases, Stabilization and Validation. The Study will collect data from multiple sites (3 to 12), and each site may enroll patients and collect data for the Stabilization and Validation Phases with a minimum of three sites for the Validation Phase.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following criteria may be enrolled in this Study:

1. Subject is male or female, age 18 or older.
2. Subject has undergone CT scan of the lung(s) that indicates one or more nodules or lesions suspicious for lung cancer.
3. Subject's pulmonary nodule or lesion is greater than 4mm. Size is determined by the largest nodule or lesion dimension identified from CT imaging.
4. Subject meets one or more of the following conditions:

   * indicated for a tissue biopsy
   * indicated for surgical resection of the lung
5. Subject must be able to receive a ProLung Test

   * within 60 days of abnormal CT (Inclusion Criterion 2 & 3)
   * within 60 days prior to the tissue biopsy or surgical resection (Inclusion Criterion 4).
6. Subject is capable of understanding and agreeing to fulfill the requirements of this Protocol.
7. Subject has signed the IRB/IEC approved Informed Consent Form ("ICF").

Exclusion Criteria

The following criteria will disqualify a subject from enrollment into this Study:

1. Subject has an implanted electronic device in the chest.
2. Subject receiving therapy for suspected chest infection such as fungal infection or tuberculosis.
3. Subject with diagnosed malignancy other than lung cancer, non-melanoma skin cancer or any cancer in which the Principal Investigator does not suspect metastatic disease to the lung, who has 2 or more suspicious pulmonary nodules.
4. Subject has received an invasive medical or surgical procedure within the thoracic cavity within 30 days prior to the ProLung Test or within the previous 14 days for a bronchoscopic procedure.
5. Subject presents with an anomalous physical or anatomical condition that precludes ProLung Test measurement.
6. Subject will have undergone unusually strenuous exercise within 24 hours.
7. Subject who has significant systemic diseases such as uncontrolled diabetes, advanced heart failure, or a recent myocardial infarction, or other medical condition such as severe morbid obesity that in the judgment of the Principal Investigator would make him/her unsuitable for the Study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with pulmonary lesions suspicious for lung cancer
Sampling Method: Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2012-10; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - UCLA Medical Center, Los Angeles, California
  - UCSD Medical Center, San Diego, California
  - Stanford University Medical Center, Stanford, California
  - Loyola University Medical Center, Maywood, Illinois
  - Greater Baltimore Medical Center, Towson, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Medical Center, Detroit, Michigan
  - University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Wake Forest University, Winston-Salem, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - Providence Health Center, Waco, Texas
  - Intermountain Healthcare, Murray, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Indeterminate Pulmonary Lesions
Started | 420
Completed | 374
Not Completed | 46

BASELINE CHARACTERISTICS:
Arm/Group | Indeterminate Pulmonary Lesions
Number analyzed (Participants) | 174
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 71
  >=65 years | 103
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92
  Male | 82
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 131
  Race: Hispanic | 15
  Race: Indian | 1
  Race: East Indian | 1
  Race: Black | 19
  Race: Asian | 6
  Race: Unkown | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinical Efficacy in the Risk Stratification of Patients With Indeterminate Lesions
Description: Demonstrate safety and efficacy in the risk stratification of patients with pulmonary lesions identified by CT that are suspicious for lung cancer.
Time Frame: The ProLung Test will be performed within 60 days of a CT Scan that identifies a lung lesion suspicious for lung cancer and evaluated once a patient diagnosis is obtained.
Population: Validation set of patients with indeterminate lung nodules
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Indeterminate Pulmonary Lesions
Number analyzed (Participants) | 174
percentage
  Positive Predictive Value | 70.37 [60.82 to 78.77]
  Negative Predictive Value | 46.97 [34.56 to 59.66]
  Sensitvity | 68.47 [58.96 to 76.96]
  Specificity | 49.21 [36.38 to 62.11]

ADVERSE EVENTS:
Time Frame: Adverse events were collected and reported on the day of measurement by the Study Device
Arm/Group | Indeterminate Pulmonary Lesions
All-Cause Mortality (participants affected / at risk) | 0/420
Serious Adverse Events (participants affected / at risk) | 0/420
Other Adverse Events (participants affected / at risk) | 3/420
OTHER ADVERSE EVENTS (reported when occurring in more than .7% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Indeterminate Pulmonary Lesions (N=420)
Discomfort at Device Measurement Location (Product Issues) | 3 (3) — 3 subjects complained of discomfort at the device measurement location on the skin. All patients who experienced an adverse event stated that they would agree to undergo measurement again.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-11-18): https://cdn.clinicaltrials.gov/large-docs/82/NCT01566682/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT01566682/SAP_001.pdf